CLINICAL TRIAL: NCT07128095
Title: COVID-19 Health Adjustments in Nutrition, General Wellness, and Exercise
Acronym: CHANGE
Status: Recruiting | Type: Observational
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Austin Robinson, Associate professor, Indiana University
Other Study IDs: IU IRB #27124
Record Dates: First submitted 2025-08-11; First posted 2025-08-17 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: COVID-19; Sleep; Immunization; Infection; Physical Inactivity; Blood Pressure; Diet Habit; Mental Health Wellness 1
Keywords: COVID-19; Sleep; Immunization; Infection; Physical Inactivity; Blood Pressure; Diet Habit; Mental Wellness
MeSH Terms: conditions — COVID-19; Infections; Sedentary Behavior; Feeding Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — During experimental visits, a blood draw will take place to assess changes in plasma electrolyte concentration, osmolality, hemoglobin, and hematocrit, and coded samples will be stored for future inflammation measures (e.g., CRP and IL-6) in addition to isolating peripheral blood mononuclear cells (PBMCs) for studying immune cell phenotype.
  Participants will also be provided with a urine collection container and corresponding form so that they can collect 24 hours of urine to enable the investigators to assess hydration biomarkers and 24-hour electrolyte (sodium, potassium, chloride) excretion, which is also used to assess dietary electrolyte intake to complement food and fluid diaries.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CHANGE participants: Male and female participants.
  Are between the ages of 18-75.
  Have a resting blood pressure no higher than 150/90 (stage 2 hypertension).
  Have a BMI below 35 kg/m2 (otherwise healthy).
  Free from metabolic disease (diabetes or renal disease), pulmonary disorders (e.g., COPD, severe asthma, and cystic fibrosis), and cardiovascular disease (peripheral vascular, cardiac, or cerebrovascular).
  Do not have any precluding medical issues that prevent participants from exercising (i.e., cardiovascular issues, or muscle/joint issues including painful arthritis) or giving blood (e.g., blood thinners).

SUMMARY:
The purpose of this study is to find out whether the COVID pandemic has affected participants' current physical activity, fitness, blood pressure, sleep, and mental stress to better understand its long-term health effects. To complete this study, participants will visit the Neurovascular Physiology Laboratory (NVPL) at the Indiana University School of Public Health Bloomington two times, requiring a total commitment of about 6 hours.

Visit 1 involves completing screening questionnaires, a consent document, and additional questionnaires about participant health behaviors (e.g., sleep and physical activity) and general mental and physical health. After the visit, participants will also start tracking their sleep and physical activity using wearable devices for 14 days, diet for at least 3 days, and blood pressure and urine for 24 hours.

Visit 2 is a second data collection visit, where participants will return the wearable devices. The investigators will measure participants' body composition, take measures of their cardiovascular health, and participants will complete a fitness test on a stationary cycle (exercise bike). The investigators will collect a 24 hour urine sample and take a blood sample to measure participants' blood glucose, electrolytes, hydration biomarkers, and markers of inflammation, as well as to study immune cells. The investigators will take participants' blood pressure at rest and during a hand-in-cold water test, which helps assess how participants' nervous system responds to stress. A full-body scan will measure participant body composition including bone density, muscle mass, and body fat percentage. Finally, participants will complete a cycling test that gradually increases in intensity to measure cardiovascular fitness.

Risks involve potential pain or bruising from blood draws, discomfort from blood pressure cuffs, stress from vigorous cycling, and psychological stress from questionnaires. There's also a slight risk of severe cardiovascular events occurring during exercise and loss of data confidentiality. Finally, the cold water test may result in a rare but noted situation where the body's nervous system overreacts to the cold stimulus, leading to a drop in blood pressure and heart rate. Participants will be monitored by trained staff during all procedures to ensure safety.

DETAILED DESCRIPTION:
The investigator will be assessing whether prior severity of COVID-19 or (Post-acute Sequelae of SARS-CoV-2 Infection) PASC is associated with reduced physical activity and cardiorespiratory fitness, impaired blood pressure regulation, worse sleep, or heightened mental stress. Participants will report to the laboratory for two visits.

Visit 1 will be comprised of participant consent, screening, and completing questionnaires surrounding sleep, stress and mental health, food security, and habitual beverage intake. Visit 1 will take approximately 2 hours in total. Participants will be asked to read the consent form at this time and be encouraged to ask any questions. Participants can then: 1) sign the consent form; 2) take it home for further consideration; or 3) decide not to participate. Participants will be screened for eligibility once written informed consent has been given. At the conclusion of the first visit, participants will be given devices to track ambulatory blood pressure for 24 hours, physical activity and sleep for ~14 days, and diet for ≥3 days (i.e., 2 week days and 1 weekend day). 24 hours before the experimental visits, participants will be given a 24-hour urine collection container to measure urine volume, urine electrolyte concentrations, urine electrolyte excretion, and urine osmolality for eventual assessment of biomarkers of kidney function and kidney injury.

Visit 2 will be an experimental visit where each participant will undergo applied physiology measures, body composition, and exercise testing. During experimental visits, a blood draw will take place to assess changes in plasma electrolyte concentration, osmolality, hemoglobin, and hematocrit, and coded samples will be stored for future inflammation measures (e.g., CRP and IL-6) in addition to isolating peripheral blood mononuclear cells (PBMCs) for studying immune cell phenotype. Participants will then have rested BP assessed. Arterial stiffness will be measured using noninvasive tonometry techniques (Pulse Wave Analysis and Pulse Wave Velocity via SphygmoCor XCEL). We will use a hand-in cold-water test (described below) to assess sympathetic nervous system excitation. The cold pressor test is where participants will submerge their hand into an ice-cold bucket of water for three minutes to elicit a sympathetic nervous system stress response. Concurrently, BP reactivity will be assessed using a cold pressor test while participants engage in submaximal exercise on a stationary bicycle. Blood pressure reactivity will be measured at the finger using a finger-specific blood pressure cuff that will measure BP on a beat-to-beat basis. A total-body dual-energy X-ray absorptiometry (iDXA) scan will be used to assess bone mineral density, lean muscle mass, fat mass, and body fat percentage. Participants will finish the visit by completing a submaximal ramp cycling test on an electronically braked cycle ergometer to assess cardiovascular fitness. The test will begin at a low workload and increase incrementally every 30 minutes until the participant reaches 70% of their estimated maximal heart rate. Heart rate, workload, and perceived exertion will be recorded throughout to estimate cardiorespiratory fitness.

Collectively, these measures will enable the investigators to determine the study objectives pertaining to whether prior COVID-19 severity or PASC impacts cardiovascular health, which have important public health implications.

ELIGIBILITY:
Inclusion Criteria:

Male and female participants. Are between the ages of 18-75. Have a resting blood pressure no higher than 150/90 (stage 2 hypertension). Have a BMI below 35 kg/m2 (otherwise healthy). Free from metabolic disease (diabetes or renal disease), pulmonary disorders (e.g., COPD, severe asthma, and cystic fibrosis), and cardiovascular disease (peripheral vascular, cardiac, or cerebrovascular).

Do not have any precluding medical issues that prevent participants from exercising (i.e., cardiovascular issues, or muscle/joint issues including painful arthritis) or giving blood (e.g., blood thinners).

Exclusion Criteria:

Younger than 18 or older than 30. Have a resting blood pressure > 150/90. Have a BMI > 35 Kg/m2 or < 18 Kg/m2. History of metabolic disease (diabetes or renal disease), pulmonary disorders (e.g., COPD, severe asthma, and cystic fibrosis), and cardiovascular disease (peripheral vascular, cardiac, or cerebrovascular).

Medical issues that prevent safe exercise (i.e., cardiovascular issues, or muscle/joint issues including painful arthritis).

Medical issues that prevent giving blood (e.g., blood thinners). Currently pregnant.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Younger than 18 or older than 75. Have a resting blood pressure > 150/90. Have a BMI > 35 Kg/m2 or < 18 Kg/m2. History of metabolic disease (diabetes or renal disease), pulmonary disorders (e.g., COPD, severe asthma, and cystic fibrosis), and cardiovascular disease (peripheral vascular, cardiac, or cerebrovascular).
  Medical issues that prevent safe exercise (i.e., cardiovascular issues, or muscle/joint issues including painful arthritis).
  Medical issues that prevent giving blood (e.g., blood thinners). Currently pregnant.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-08-22 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Brachial blood pressure | Through study completion (two-1.5 hour study visits)
  Seated rachial blood pressure will be measured triplicate after at least 5 minutes of rest using an oscillometric device (Suntech CT 40)
24-hour ambulatory blood pressure | During the second data collection visit
  Participants will wear an Oscar2 (with SphygmoCor) ambulatory blood pressure monitor on their upper arm for up to 24-hours after their second study visit to measure systolic and diastolic blood pressure. The purpose of the ambulatory blood pressure monitoring is to determine blood pressure regulation over an entire day. This blood pressure monitor will be set to automatically take blood pressure every 20 minutes. The monitor records and saves each blood pressure measurement automatically.

SECONDARY OUTCOMES:
Objective sleep duration | 14 days
  LEAP ActiWatch will be used to quantify sleep duration in hours. Participants will wear the watch units for 14 days. The investigators will assess sleep duration and cross-check actigraphy wear times with a sleep diary.
Objective sleep efficiency | 14 days
  LEAP ActiWatch will be used to quantify the percentage of time in bed actually spent sleeping to calculate sleep efficiency.
Subjective sleep duration | 14 days
  Sleep quality and disturbances will be evaluated using validated self-reported questionnaires, including the Pittsburgh Sleep Quality Index (PSQI), Munich Sleep Questionnaire (MCQ), Insomnia Severity Index (ISI), and an obstructive sleep apnea scale (i.e., STOP-BANG).
  The investigators will use the Pittsburgh Sleep Quality Index (PSQI) to assess sleep duration reflective of the one-month period leading into the study. This outcome is specifically referring to self-reported sleep duration in hours.
Subjective sleep quality | 14 days
  The Pittsburgh Sleep Quality Index (PSQI) will assess perceived sleep quality reflective of the one-month period leading into the study. The Insomnia Severity Index, the Munich Sleep Questionnaire, and the Obstructive Sleep Apnea Scale will additionally measure sleep quality.
Diet quality | Measured at baseline
  Diet will be measured by the Nutrition Data System for Research software. We will obtain macronutrients, micronutrients, and the Healthy Eating Index

OTHER OUTCOMES:
Perceived stress | Measured at baseline
  We will measure perceived stress (using the Perceived Stress Scale) and stress coping ability using the Connor-Davidson Resilience Scale
Blood pressure reactivity | Measured for 3 minutes during the second data collection visit
  Blood pressure reactivity (via the cold pressor test)
Inflammatory markers | Measured during the second data collection visit
  Circulating immune cells and inflammatory markers, such as C-reactive protein (CRP), interleukin-6 (IL-6), and potentially other cytokines, will be quantified using blood samples.
Hope | Measured at baseline
  Measured using adult hope scale. The scale is a 12-item questionnaire measuring an individual's level of hope, where I higher score indicates greater hope.
Mood | Measured at baseline
  Profile of Mood States is a psychological rating scale used to measure six identifiable mood or affective states: Tension-Anxiety, Depression-Dejection, Anger-Hostility, Vigor-Activity, Fatigue-Inertia, and Confusion-Bewilderment. It is a 65 item scale, using a 5 point scale for each item. 0="Not at all", 4="Extremely".

CONTACTS AND LOCATIONS:
Overall Officials: Austin T Robinson, PhD, Principal Investigator — Indiana University
Locations (1):
- Indiana University School of Public Health, Bloomington, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
Unidentified individual participant data will be made available to other researchers upon reasonable request and data and material transfer agreement
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: 2 years after completion of the study, indefinitely
Access Criteria: Unidentified individual participant data will be made available to other researchers upon reasonable request and data and completion of a material transfer agreement with Indiana University.